CLINICAL TRIAL: NCT07324746
Title: Effectiveness of a Herbal Supplement Containing Boswellia Serrata, Curcuma Longa, and Vitis Vinifera in Patients With Osteoarthritis.
Brief Title: The Effectiveness of a Herbal Supplement in Osteoarthritis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Middlesex University (Other)
Responsible Party: Principal Investigator, Patrycja Brodka Pedro, PhD Student in Biomedicine, Bioscience Laboratory Technician, Middlesex University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 30400
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis (OA); Osteoarthritis (OA) of the Hip; Osteoarthritis (OA) of the Knee; Osteoarthritis
Keywords: Boswellia serrata; Curcuma longa; Curcumin; Turmeric; Osteoarthritis; Grape extract; Knee osteoarthritis; Hip osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: A randomised, double-blind, crossover study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): Dietary supplement containing standardised herbal extracts of Boswellia Serrata (525 mg), Curcuma Longa (150 mg), Vitis vinifera (75 mg)
  Interventions: Dietary Supplement: Active treatment
- Placebo (Placebo Comparator): Dietary supplement placebo containing no standardised herbal extracts or other active ingredients.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Active treatment — A dietary supplement containing standardised herbal extracts of Boswellia serrata (525 mg), Curcuma longa (150 mg), Vitis vinifera (75 mg). Four times a day.
  Arms: Active Treatment
Other: Placebo — A placebo containing no standardised herbal extracts or other active ingredients. Four times a day.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effectiveness and safety of a combined herbal supplement containing Boswellia serrata, Curcuma longa, and Vitis vinifera in adults with clinically diagnosed knee or hip osteoarthritis.

The primary objective is to determine whether the supplement improves osteoarthritis-related symptoms.

The supplement will be compared with a placebo.

Participants will:

* take the supplement and placebo for 4 weeks each, one at a time;
* complete validated questionnaires (6 times online)
* perform three performance-based physical tests (6 times online)
* provide a urine sample

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18
* Diagnosis of osteoarthritis in knee or hip
* Numerical Rating Scale (NRS) ≥ 4 during the most painful movement in the last 24 hours
* Lequesne's Functional Index (LFI) score ≥ 7
* Ambulant patient

Exclusion Criteria:

* Pregnant and breastfeeding
* Autoimmune disease such as rheumatoid arthritis, gout, lupus
* Joint trauma, joint injury, joint infection, meniscus tear, complete loss of articular cartilage
* Expectation of surgery
* History of the viscous or corticosteroids injections into affected joints or oral corticosteroids within last 12 months
* Allergy to one of the intervention's ingredients or NSAIDs
* Peptic ulceration and upper gastrointestinal haemorrhage
* High alcohol intake, inability to abstain from alcohol, substance abuse, history of addiction
* Tumor, cancer
* Abnormal renal or/and hepatic functions or altered blood chemistry
* Use of concomitant medication able to interfere with the interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) score | Change from the start of the intervention to Week 4 of supplementation
  Western Ontario and McMaster Universities Arthritis Index, a validated, specialised instrument used to assess pain, stiffness, and physical function in people with osteoarthritis. Scores range from 0 to 96 (Likert version), with higher scores indicating worse pain (0-20), stiffness (0-8), and physical function (0-68).
Change in Numeric Rating Scale (NRS) score | Change from the start of the intervention to Week 4 of supplementation
  Numeric Rating Scale. A specialised pain assessment tool, where patients rate their pain intensity on a scale from 0 to 10, where 0 indicates no pain and 10 indicates worst imaginable pain; higher scores indicate worse outcomes.
Change in Intermittent and Constant Osteoarthritis Pain knee/hip (ICOAP) score | Change from the start of the intervention to Week 4 of supplementation
  ICOAP. A Measure of Intermittent and Constant Osteoarthritis Pain knee/hip To assess two distinct types of pain experienced by people with osteoarthritis-intermittent pain (comes and goes, 0 - 24) and constant pain (persistent, ongoing pain, 0 - 20). Scores range from 0 to 44, with higher scores indicating more severe osteoarthritis related pain.
Change in EuroQol 5-Dimension 5-Level (EQ-5D-5L) score | Change from the start of the intervention to Week 4 of supplementation
  EuroQol 5-Dimension 5-Level questionnaire. A generic, widely used tool to measure health-related quality of life. It measures five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression. A score of 1 indicates no problems, while 5 indicates extreme problems in the respective dimension.
  In addition, the EQ Visual Analogue Scale (EQ-VAS) records the respondent's self-rated health on a vertical scale ranging from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Change in urinary C-terminal telopeptide of type II collagen (uCTX-II) levels | Change from the start of the intervention to Week 4 of supplementation
  uCTX-II (urinary C-terminal telopeptide of type II collagen) is a biochemical marker measured in urine that reflects type II collagen degradation, which occurs primarily in articular cartilage.

SECONDARY OUTCOMES:
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) score. | Change from baseline to the end of Week 1 of supplementation
  Western Ontario and McMaster Universities Arthritis Index, a validated, specialised instrument used to assess pain, stiffness, and physical function in people with osteoarthritis. Scores range from 0 to 96 (Likert version), with higher scores indicating worse pain (0-20), stiffness (0-8), and physical function (0-68).
Change in Numeric Rating Scale (NRS) score | Change from baseline to the end of Week 1 of supplementation
  Numeric Rating Scale. A specialised pain assessment tool, where patients rate their pain intensity on a scale from 0 to 10, where 0 indicates no pain and 10 indicates worst imaginable pain; higher scores indicate worse outcomes.
Change in Intermittent and Constant Osteoarthritis Pain knee/hip (ICOAP) score | Change from baseline to the end of Week 1 of supplementation
  ICOAP. A Measure of Intermittent and Constant Osteoarthritis Pain knee/hip To assess two distinct types of pain experienced by people with osteoarthritis-intermittent pain (comes and goes, 0 - 24) and constant pain (persistent, ongoing pain, 0 - 20). Scores range from 0 to 44, with higher scores indicating more severe osteoarthritis related pain.
Change in Lequesne Functional Index (LFI) score | Change from baseline to the end of Week 1 of supplementation
  Lequesne Functional Index. A specialised questionnaire used to evaluate the severity of osteoarthritis and its impact on daily function, particularly for the hip and knee. Scores range from 0 to 24, with higher scores indicating greater severity and worse functional impairment.
Change in Lequesne Functional Index (LFI) score | Change from the start of the intervention to Week 4 of supplementation
  Lequesne Functional Index. A specialised questionnaire used to evaluate the severity of osteoarthritis and its impact on daily function, particularly for the hip and knee. Scores range from 0 to 24, with higher scores indicating greater severity and worse functional impairment.
Evaluation of Minimal Clinically Important Difference for measured scores | Change from the start of the intervention to Week 4 of supplementation
  Minimal Clinically Important Difference assessed by Patient Global Impression of Change.
  PGIC is a specialised patient-reported outcome tool.
Change in 30-Second Chair Stand Test | Change from baseline to the end of Week 1 of supplementation
  30-Second Chair Stand Test is a functional assessment that measures lower-body strength and endurance by recording the number of times an individual can rise to a full standing position from a seated position in 30 seconds, without using their arms.
Change in 30-Second Chair Stand Test | Change from the start of the intervention to Week 4 of supplementation
  30-Second Chair Stand Test is a functional assessment that measures lower-body strength and endurance by recording the number of times an individual can rise to a full standing position from a seated position in 30 seconds, without using their arms.
Change in Stair Climb Test | Change from baseline to the end of Week 1 of supplementation
  Stair Climb Test is a functional performance assessment that measures lower-limb strength, power, and mobility by timing how quickly an individual ascends and descends a set of stairs.
Change in Stair Climb Test | Change from the start of the intervention to Week 4 of supplementation
  Stair Climb Test is a functional performance assessment that measures lower-limb strength, power, and mobility by timing how quickly an individual ascends and descends a set of stairs.
Change in 40-metre Fast-Paced Walk Test | Change from baseline to the end of Week 1 of supplementation
  The 40-metre Fast-Paced Walk Test (4 × 10 m) is a functional mobility assessment that measures walking speed and dynamic balance by timing how quickly an individual completes four 10-metre walks at a fast but safe pace.
Change in the 40-metre Fast-Paced Walk Test (4 × 10 m) | Change from the start of the intervention to Week 4 of supplementation
  The 40-metre Fast-Paced Walk Test (4 × 10 m) is a functional mobility assessment that measures walking speed and dynamic balance by timing how quickly an individual completes four 10-metre walks at a fast but safe pace.
Global Physical Activity Questionnaire | Change from the start of the intervention to Week 4 of supplementation
  The GPAQ will be used to monitor physical activity patterns in participants, and detect possible changes.
Adverse events | The length of intervention: 4 weeks
  Collection of adverse events to assess the safety and tolerability of the supplement
Rescue medication | The length of intervention: 4 weeks
  The use of rescue medication

OTHER OUTCOMES:
Satisfaction with remotely controlled study | At the end of the study: 12 weeks
  Participants will be asked to complete a remote study satisfaction survey

CONTACTS AND LOCATIONS:
Locations (1):
- Middlesex Univeristy London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No